CLINICAL TRIAL: NCT05706519
Title: Metabolomics, Genomics and Nutrition for Cardiovascular Disease Precision Medicine
Acronym: OMIC-CARD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Other Study IDs: PMP21/00125
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Heart Disease; Coronary Heart Disease
Keywords: Metabolomics; Mediterranean Diet; Ischemic Heart Disease; Food Patterns; Dietary Assessment Methods
MeSH Terms: conditions — Myocardial Ischemia; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — The Biospecimen sample for this study will be the blood draw of serum and plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Six hundred volunteers. This group has to be without any type of cardiovascular Disease.
- Case Group: Six hundred volunteers. In this group, participants must present a diagnosis of ischemic heart disease at least 1 year but less than 5 years from recruitment

SUMMARY:
The objective of this project is to validate, through high-throughput advanced metabolomics techniques, the nutritional assessment tools to be used in the IMPaCT cohort. At the same time, the ability of metabolomics fingerprints of nutritional patterns to discriminate between patients with and without major cardiovascular disease will be identified. Finally, the modification of these predictions will be evaluated based on the genetic profiles. The main hypothesis holds that the integration of metabolomics, genomic and nutritional information will serve to personalize the approach to cardiovascular disease, both in prevention and treatment, and that these tools, in turn, will be valid enough to be applied systematically and efficiently in the IMPaCT cohort.

DETAILED DESCRIPTION:
In two independent samples, one of 600 subjects free of cardiovascular disease (control group) and the other of 600 subjects with a history of ischemic heart disease (established heart disease group) eating habits will be evaluated using Food Frequency Questionnaire, based on those repeatedly used in epidemiological studies carried out in Spain, as well as other nutritional evaluation tools. Each participant will undergo a complete plasma metabolomics profile with identification of > 300 metabolites and a complete genome-wide association analysis. Artificial intelligence models and elastic net regression self-learning algorithms will be applied to select the metabolomics fingerprint of eating patterns.

The objectives are:

* To assess whether the relationship between diet and metabolic footprint is similar in those with established Cardio Vascular Disease or not. This will allow evaluating the usefulness of metabolic fingerprint to monitor the metabolic response to diet in patients with Cardio Vascular Disease and thus help to individualize their pharmacological and non-pharmacological treatment (diet and lifestyle)
* If there are sociodemographic characteristics - including the gender perspective-, clinical or genetic characteristics that help identify people who present a greater metabolic response to diet both in people without and in people with Cardio Vascular Disease.
* If the possible limitations of the metabolic footprint of different dietary patterns are reduced by using different tools for the collection of nutritional information. Self -completed Food Frequency Questionnaire a, Food Frequency Questionnaire b completed with telephone interviewer, brief assessment tools, and 4 dietary records of 3 days each distributed throughout the year will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 - 79 years old
* Living in Spain for more than 2 years
* Fluent in Spanish
* Ability for answer all the study questionaries'
* Ability to validly grant informed consent
* Ability to move on one's own
* Not under palliative care due to serious illness, institutionalized population will not be recruited
* Not planning any change of address to another autonomous community within a year.
* Receive health care in National Health System. Officials or self-employed workers with health coverage exclusively in "Mutuas" that do not allow telematics access to health data will be excluded.

Exclusion Criteria:

* Chronic alcoholism or regular alcohol consumption > 80 g/d
* BMI >40 kg/m²
* Participation in a clinical trial conducted with drugs or use of any drug in experimental status during the year prior to inclusion
* Patient with cancer treatment two years before
* Patient with history of gastrectomy or intestinal resection. Patients with acute infection or inflammatory process (e.g. Pneumonia), may be included in the study three months after the infectious process.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Six recruitment nodes were established, each one from a different Autonomous Community (Andalusia, Cantabria, The Balearic Islands, Madrid, Navarra, and the Basque Country), Comprising cardiologist and primary care clinicians. In each of the 6 nodes, 100 participants without ischemic heart disease (ICD) will be recruited for the control group and another 100 for the case group. The controls will be selected through the health Centers, The cases will be selected in CS and in Cardiology consultations of the National Health Service (NHS).
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Metabolomics | Baseline
  Human plasma and serum will be analysed to obtain chemical information of the different families of metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Buil- Cosiales, Doctor, Principal Investigator — Servicio Navarro de Salud - Osasunbidea
Locations (6):
- Spain (6):
  - ibs.GRANADA, Granada, Andalusia
  - Instituto de Investigación Sanitaria, Vitoria-Gasteiz, Araba
  - Institut D' Investigació Sanitària Illes Balears, Palma de Mallorca, Balearic Islands
  - Universidad de Cantabria, Santander, Cantabria
  - Servicio Navarro de Salud Osasunbidea, Pamplona, Navarre
  - UAM, Madrid